CLINICAL TRIAL: NCT00469560
Title: Open Label, Multicenter Study to Evaluate Safety/Tolerability and Efficacy of Deferasirox (ICL670) in Myelodysplastic Syndrome Patients With Chronic Transfusional Hemosiderosis.
Brief Title: Safety, Tolerability, and Efficacy of Deferasirox in MDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDS0306
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Myelodysplastic Syndromes; Hemosiderosis
Keywords: MDS; Chronic transfusional hemosiderosis; Deferasirox
MeSH Terms: conditions — Myelodysplastic Syndromes; Hemosiderosis | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox (Experimental)
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox

SUMMARY:
Open label, single arm study on Deferasirox treatment in MDS patients with chronic transfusional hemosiderosis.

Patients receive daily oral dosis of Deferasirox in order to eliminate the quantity of iron administered during transfusions and, if needed, to reduce the overload of already present iron.

After an screening phase in which patients are evaluated according to eligibility criteria, a one year treatment phase foresees monthly visits to evaluate safety and efficacy signs.

DETAILED DESCRIPTION:
It has been widely shown that an appropriate chelating therapy in chronic anemias transfusion dependent can prevent the overstock of iron and can reduce the already existing overstock reducing, then, the co-morbidity and improving survival.

In particular, some authors have shown in MDS affected patients undergoing intensive chelating therapy with deferoxamine haematological recovery with a reduction of the need of transfusions.

With the present study, we plan to evaluate the safety and efficacy of a therapy with the new oral chelating Deferasirox in MDS patients with transfusional hemosiderosis.

This is an open label, single arm study on Deferasirox treatment in MDS patients with chronic transfusional hemosiderosis.

Patients will receive daily oral dosis of Deferasirox in order to eliminate the quantity of iron administered during transfusions and, if needed, to reduce the overload of already present iron.

After an screening phase in which patients are evaluated according to eligibility criteria, a one year treatment phase foresees monthly visits to evaluate safety and efficacy signs.

ELIGIBILITY:
Inclusion Criteria:

* Patients, both males and females, with low and intermediate I risk (IPSS score) Myelodysplastic syndrome and transfusion-induced hemosiderosis.
* Age >=18 years
* Patients who never received chelation therapy or who received a therapy with Desferal after a day of wash out
* Medical history of at least 20 blood transfusions (equivalent to 100 ml/kg of red cells concentrate).
* Availability of data concerning blood transfusions during the 12 weeks before screening
* Serum ferritin >= 1000 µg/L at least twice (at least 2 week interval between the 2 analysis) during the year before the screening
* Life expectancy > 12 months
* Availability of at least 3 complete blood counts (before transfusions) during the 12 weeks before the screening

Exclusion Criteria:

* Diagnosis different from MDS (i.e. myelofibrosis)
* Severe renal impairment (creatinine clearance < 60 ml/min)
* ALT/AST > 500 U/L
* Active B and/or C hepatitis
* Patients treated during the past 4 weeks with experimental drugs for MDS (including thalidomide, azacitidine, arsenic trioxide). These patients become eligible after a "wash out" of at least 4 weeks
* Concomitant treatment with another iron-chelating agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the tolerability and safety profile of Deferasirox in pts with MDS with post-transfusional hemosiderosis | On a monthly basis thereafter from baseline assessment.

SECONDARY OUTCOMES:
To evaluate Deferasirox efficacy as chelation therapy in terms of reduction of serum ferritin levels compared to basal levels | At 3, 6, 9, and 12 months from baseline assessment.
To evaluate the impact Deferasirox iron chelating therapy vs the normal demand of transfusions in a subgroup of pts that will not receive growth factors or chemotherapy according to their basal characteristics. | On a monthly basis thereafter from baseline assessment.
Quality of Life evaluation. | At 3, 6, 9, and 12 months from baseline assessment.
Compliance to chelating therapy evaluation. | On a monthly basis thereafter from baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele ANGELUCCI, Pr., Principal Investigator — Ospedale "A. Businco", Cagliari
Locations (17):
- Italy (17):
  - SOC EMATOLOGIA ASO SS Antonio e Biagio, Alessandria
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna
  - CTMO-Ematologia Ospedale Binaghi, Cagliari
  - Ospedale "A. Businco", Cagliari
  - Oncoematologia "A.O.R.N. S'Anna e S.Sebastiano", Caserta
  - US Dipartimentale Centro per le Malattie del Sangue, Castelfranco Veneto
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Policlinico di Careggi, Università delgi studi di Firenze, Florence
  - Clinica Ematologica - Università degli Studi, Genova
  - Divisione di Ematologia e TMO - Ospedale "A. Cardarelli "- Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Clinica Ematol Università di Perugia, Policlinico Monteluce, Perugia
  - Ematologia- Università degli Studi "La Sapienza", Roma
  - Università Cattolica del Sacro Cuore, Roma
  - Università degli Studi di Tor Vergata, Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - Ospedale Civile SS. Giovanni e Paolo, Venezia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Alessandrino EP, Amadori S, Barosi G, Cazzola M, Grossi A, Liberato LN, Locatelli F, Marchetti M, Morra E, Rebulla P, Visani G, Tura S; Italian Society of Hematology. Evidence- and consensus-based practice guidelines for the therapy of primary myelodysplastic syndromes. A statement from the Italian Society of Hematology. Haematologica. 2002 Dec;87(12):1286-306. PMID 12495903
- [Background] Anderson LJ, Holden S, Davis B, Prescott E, Charrier CC, Bunce NH, Firmin DN, Wonke B, Porter J, Walker JM, Pennell DJ. Cardiovascular T2-star (T2*) magnetic resonance for the early diagnosis of myocardial iron overload. Eur Heart J. 2001 Dec;22(23):2171-9. doi: 10.1053/euhj.2001.2822. PMID 11913479
- [Background] Borgna-Pignatti C, Franchini M, Gandini G, Vassanelli A, De Gironcoli M, Aprili G. Subcutaneous bolus injection of deferoxamine in adult patients affected by onco-hematologic diseases and iron overload. Haematologica. 1998 Sep;83(9):788-90. PMID 9825575
- [Background] Efficace F, Bottomley A, Osoba D, Gotay C, Flechtner H, D'haese S, Zurlo A. Beyond the development of health-related quality-of-life (HRQOL) measures: a checklist for evaluating HRQOL outcomes in cancer clinical trials--does HRQOL evaluation in prostate cancer research inform clinical decision making? J Clin Oncol. 2003 Sep 15;21(18):3502-11. doi: 10.1200/JCO.2003.12.121. PMID 12972527
- [Background] Caocci G, Baccoli R, Ledda A, Littera R, La Nasa G. A mathematical model for the evaluation of amplitude of hemoglobin fluctuations in elderly anemic patients affected by myelodysplastic syndromes: correlation with quality of life and fatigue. Leuk Res. 2007 Feb;31(2):249-52. doi: 10.1016/j.leukres.2006.05.015. Epub 2006 Jun 30. PMID 16814382
- [Background] Galanello R. Evaluation of ICL670, a once-daily oral iron chelator in a phase III clinical trial of beta-thalassemia patients with transfusional iron overload. Ann N Y Acad Sci. 2005;1054:183-5. doi: 10.1196/annals.1345.021. PMID 16339664
- [Derived] Efficace F, Santini V, La Nasa G, Cottone F, Finelli C, Borin L, Quaresmini G, Di Tucci AA, Volpe A, Cilloni D, Quarta G, Sanpaolo G, Rivellini F, Salvi F, Molteni A, Voso MT, Alimena G, Fenu S, Mandelli F, Angelucci E. Health-related quality of life in transfusion-dependent patients with myelodysplastic syndromes: a prospective study to assess the impact of iron chelation therapy. BMJ Support Palliat Care. 2016 Mar;6(1):80-8. doi: 10.1136/bmjspcare-2014-000726. Epub 2014 Sep 9. PMID 25204541